CLINICAL TRIAL: NCT02434328
Title: A Two-year, Randomized, Double-masked, Multicenter, Two-arm Study Comparing the Efficacy and Safety of RTH258 6 mg Versus Aflibercept in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: Efficacy and Safety of RTH258 Versus Aflibercept - Study 2
Acronym: HARRIER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTH258-C002; 2014-004886-26 (EudraCT Number); CRTH258A2302 (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2015-03-27; First posted 2015-05-05 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Neovascular Age-Related Macular Degeneration; Choroidal Neovascularization
Keywords: AMD; CNV; IVT
MeSH Terms: conditions — Choroidal Neovascularization | interventions — brolucizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brolucizumab 6 mg (Experimental): Single intravitreal (IVT) injection of brolucizumab at Day 0, Week 4, and Week 8, followed by 1 injection every 8 weeks/1 injection every 12 weeks (q8w/q12w) maintenance regimen until study exit
  Interventions: Drug: Brolucizumab ophthalmic solution
- Aflibercept 2 mg (Active Comparator): Single IVT injection of aflibercept ophthalmic solution at Day 0, Week 4, and Week 8, followed by q8w maintenance regimen until study exit
  Interventions: Drug: Aflibercept ophthalmic solution

INTERVENTIONS:
Drug: Brolucizumab ophthalmic solution — Ophthalmic solution for IVT injection administered as a 6 mg/50 µL dose
  Other Names: RTH258
  Arms: Brolucizumab 6 mg
Drug: Aflibercept ophthalmic solution — Ophthalmic solution for IVT injection administered as a 2 mg/50 µL dose
  Other Names: EYLEA®
  Arms: Aflibercept 2 mg

SUMMARY:
The purpose of this study is to compare brolucizumab (RTH258) ophthalmic solution for intravitreal (IVT) injection (6 mg) to aflibercept ophthalmic solution for IVT injection (2 mg) in subjects with untreated active choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD) in the study eye.

DETAILED DESCRIPTION:
Subjects were randomized to brolucizumab 6 mg and aflibercept 2 mg in a 1:1 ratio. Subjects in both treatment arms received 3 monthly loading doses (Day 0, Week 4 and Week 8), followed by a maintenance regimen, until the end of the study (Week 96/Exit). All subjects attended pre-specified visits every 4 weeks.

Subjects in the brolucizumab 6 mg arm followed a q12w/q8w maintenance regimen. Within the q12w/q8w regimen, the initial treatment after the loading phase was q12w (1 injection every 12 weeks). If disease activity was identified by the masked investigator at any of the disease activity assessments, dosing was adjusted to q8w (1 injection every 8 weeks) ("q12w/q8w regimen"). Once subjects were adjusted to the q8w interval, they stayed on that interval until the end of the study.

Subjects in the aflibercept 2 mg arm followed a q8w maintenance regimen until the end of the study.

Results reported up to Week 48 are based on the database locked for the primary analysis at Week 48. Results reported after Week 48 are based on the database locked at the end of study (final analysis).

ELIGIBILITY:
Key Inclusion Criteria:

* Provide written informed consent;
* Active CNV lesions secondary to AMD that affected the central subfield in the study eye at Screening;
* Total area of CNV > 50% of the total lesion area in the study eye at Screening;
* Intraretinal and/or subretinal fluid affecting the central subfield of the study eye at Screening;
* Best corrected visual acuity (BCVA) between 78 and 23 letters, inclusive, in the study eye at Screening and Baseline using Early Treatment Diabetic Retinopathy Study (ETDRS) testing.

Key Exclusion Criteria:

* Any active intraocular or periocular infection or active intraocular inflammation in either eye at Baseline;
* Central subfield of the study eye affected by fibrosis or geographic atrophy or total area of fibrosis ≥ 50% of the total lesion in the study eye at Screening;
* Subretinal blood affecting the foveal center point and/or ≥ 50% of the lesion of the study eye at Screening;
* Any approved or investigational treatment for neovascular age-related macular degeneration (nAMD) in the study eye at any time;
* Retinal pigment epithelial rip/tear in the study eye at Screening or Baseline or current vitreous hemorrhage or history of vitreous hemorrhage in the study eye within 4 weeks prior to Baseline;
* Pregnant or nursing women; women of child-bearing potential;
* Stroke or myocardial infarction in the 6-month period prior to Baseline.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1048 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2018-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Group Trial Lead, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Khanani AM, Sadda SR, Sarraf D, Tadayoni R, Wong DT, Kempf AS, Saffar I, Gedif K, Chang A. Effect of Brolucizumab and Aflibercept on the Maximum Thickness of Pigment Epithelial Detachments and Sub-Retinal Pigment Epithelium Fluid in HAWK and HARRIER. Ophthalmol Retina. 2025 Jan;9(1):13-21. doi: 10.1016/j.oret.2024.07.012. Epub 2024 Jul 19. PMID 39033924
- [Derived] Singh RP, Jhaveri C, Wykoff CC, Gale RP, Staurenghi G, Iida T, Koh A, B G, Gedif K, Singer M. Efficacy Outcomes of Brolucizumab Versus Aflibercept in Neovascular Age-Related Macular Degeneration Patients with Early Residual Fluid. Ophthalmol Retina. 2022 May;6(5):377-386. doi: 10.1016/j.oret.2021.12.014. Epub 2021 Dec 27. PMID 34968756
- [Derived] Mones J, Srivastava SK, Jaffe GJ, Tadayoni R, Albini TA, Kaiser PK, Holz FG, Korobelnik JF, Kim IK, Pruente C, Murray TG, Heier JS. Risk of Inflammation, Retinal Vasculitis, and Retinal Occlusion-Related Events with Brolucizumab: Post Hoc Review of HAWK and HARRIER. Ophthalmology. 2021 Jul;128(7):1050-1059. doi: 10.1016/j.ophtha.2020.11.011. Epub 2020 Nov 15. PMID 33207259
- [Derived] Dugel PU, Koh A, Ogura Y, Jaffe GJ, Schmidt-Erfurth U, Brown DM, Gomes AV, Warburton J, Weichselberger A, Holz FG; HAWK and HARRIER Study Investigators. HAWK and HARRIER: Phase 3, Multicenter, Randomized, Double-Masked Trials of Brolucizumab for Neovascular Age-Related Macular Degeneration. Ophthalmology. 2020 Jan;127(1):72-84. doi: 10.1016/j.ophtha.2019.04.017. Epub 2019 Apr 12. PMID 30986442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from investigative sites located in Austria, Belgium, Croatia, Czech Republic, Denmark, Estonia, Finland, France, Germany, Greece, Hungary, Ireland, Italy, South Korea, Latvia, Lithuania, Netherlands, Norway, Poland, Portugal, Russia, Singapore, Slovakia, Spain, Switzerland, Taiwan, Turkey, UK, and Vietnam.
Pre-assignment Details: Of the 1048 subjects enrolled in the study, 305 were exited prior to randomization as screen failures. This reporting group includes all randomized subjects.
Groups:
- Aflibercept 2 mg: Single IVT injection of aflibercept at Day 0, Week 4, and Week 8, followed by q8w maintenance regimen until study exit
Period: Overall Study
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Started (All randomized subjects) | 372 | 371
Randomized and Treated | 370 | 369
Completed | 342 | 329
Not Completed | 30 | 42
Not completed — Adverse Event | 9 | 4
Not completed — Lack of Efficacy | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 12 | 21
Not completed — Death | 4 | 7
Not completed — Lost to Follow-up | 1 | 6
Not completed — Other | 4 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who received at least 1 IVT injection of study treatment (Full Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg | Total
Number analyzed (Participants) | 370 | 369 | 739
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (8.58) | 75.5 (7.87) | 75.1 (8.24)
Age, Customized [Number; unit: participants]
  less than 50 years | 0 | 0 | 0
  50-64 years | 44 | 28 | 72
  65-74 years | 124 | 126 | 250
  75-84 years | 150 | 167 | 317
  85 years and greater | 52 | 48 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 212 | 422
  Male | 160 | 157 | 317
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 25 | 48
  Not Hispanic or Latino | 321 | 322 | 643
  Unknown or Not Reported | 26 | 22 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 23 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 340 | 341 | 681
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 5 | 4 | 9
Best Corrected Visual Acuity (BCVA) (letters read) [Mean (Standard Deviation); unit: letters] — BCVA (with spectacles or other visual corrective devices) was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) testing at 4 meters and reported in letters read correctly. Baseline was defined as the last measurement prior to first treatment. An increase (gain) in letters read from the baseline assessment indicates improvement. One eye (study eye) contributed to the analysis.
  letters | 61.5 (12.59) | 60.8 (12.93) | 61.2 (12.76)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) (Letters Read) at Week 48 - Study Eye
Description: BCVA (with spectacles or other visual corrective devices) was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) testing at 4 meters and reported in letters read correctly. Baseline was defined as the last measurement prior to first treatment. An increase (gain) in letters read from the baseline assessment indicates improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 48
Population: Full Analysis Set (FAS) - Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: letters
Groups:
- Brolucizumab 6 mg: Single IVT injection of brolucizumab at Day 0, Week 4, and Week 8, followed by q8w/q12w maintenance regimen until study exit
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
letters | 6.9 (11.47) | 7.6 (12.47)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Non-Inferiority — The noninferiority margin was 4 letters; p < 0.0001, ANOVA — 1-sided p-value reported. Hypothesis tested according to the pre-specified hierarchical testing that ensures the global type I error rate at 0.05; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-2.4 to 1.0], Standard Error of Mean 0.86 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

2. Secondary Outcome: Average Change From Baseline in BCVA (Letters Read) Over the Period Week 36 Through Week 48 - Study Eye
Description: BCVA (with spectacles or other visual corrective devices) was assessed using ETDRS testing at 4 meters and reported in letters read correctly. For each subject, this endpoint was defined as the average of the changes from baseline to Weeks 36, 40, 44, and 48. Baseline was defined as the last measurement prior to first treatment. An increase (gain) in letters read from the baseline assessment indicates improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Weeks 36, 40, 44, 48
Population: FAS - LOCF
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
letters | 6.6 (11.10) | 7.7 (11.81)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Non-Inferiority — The non-inferiority margin was 4 letters; p = 0.0003, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -1.2, 95% CI 2-sided [-2.8 to 0.5], Standard Error of Mean 0.82 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

3. Secondary Outcome: Proportion of Subjects With Positive q12 (Every 12 Weeks) Treatment Status at Week 48
Description: Positive q12 treatment status was defined as IVT injections per planned dosing regimen (one injection every 12 weeks "q12w", after the initial three loading injections every 4 weeks "q4w"). A disease activity assessment (DAA) was performed at pre-specified visits (Weeks 16, 20, 28, 32, 40, 44) to identify q8w (one injection every 8 weeks) need. The estimate for the proportion of subjects with a positive q12w status at Week 48 were derived from Kaplan-Meier time to event analyses for the event of first q8w need, applying event allocations (in case of lack of efficacy and/or lack of safety=efficacy/safety approach) and censoring as described in the SAP. Censored subjects were considered to be not anymore under risk for a q8 need identification at later visits. Corresponding 95% Confidence Intervals (CIs) were derived from the LOGLOG transformation. This outcome measure was pre-specified for brolucizumab 6 mg arm only. Hypothesis testing not pre-specified.
Time Frame: Weeks 16, 20, 28, 32, 40, 44, 48
Population: FAS - efficacy/safety approach
Measure: Number (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 370
proportion of subjects | 0.5101 [0.4567 to 0.5610]

4. Secondary Outcome: Proportion of Subjects With Positive q12 Treatment Status at Week 48 Within the Subjects With no q8 (Every 8 Weeks) Treatment Need During the Initial q12w Cycle (Week 16, Week 20)
Description: Positive q12 treatment status was defined as IVT injections per planned dosing regimen (one injection every 12 weeks "q12w", after the initial three loading injections every 4 weeks "q4w"). A disease activity assessment (DAA) was performed at pre-specified visits (Weeks 16, 20, 28, 32, 40, 44) to identify q8w need. The estimate for the proportion of subjects with a positive q12w status at Week 48 were derived from Kaplan-Meier time to event analyses for the event of first q8w need, applying event allocations (in case of lack of efficacy and/or lack of safety=efficacy/safety approach) and censoring as described in the SAP. Censored subjects were considered to be not anymore under risk for a q8 need identification at later visits. Corresponding 95% Confidence Intervals (CIs) were derived from the LOGLOG transformation. This outcome measure was pre-specified for brolucizumab 6 mg arm only. Hypothesis testing not pre-specified.
Time Frame: Weeks 16, 20, 28, 32, 40, 44, 48
Population: FAS - efficacy/safety approach
Measure: Number (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 220
proportion of subjects | 0.8170 [0.7582 to 0.8629]

5. Secondary Outcome: Proportion of Subjects With Positive q12 Treatment Status up to Week 96
Description: Positive q12 treatment status was defined as IVT injections per planned dosing regimen (one injection every 12 weeks "q12w", after the initial three loading injections every 4 weeks "q4w"). A disease activity assessment (DAA) was performed at pre-specified visits (Weeks 16, 20, 28, 32, 40, 44, 52, 56, 64, 68, 76, 80, 88, 92) to identify q8w need. The estimate for the proportion of subjects with a positive q12w status at Week 48 were derived from Kaplan-Meier time to event analyses for the event of first q8w need, applying event allocations (in case of lack of efficacy and/or lack of safety=efficacy/safety approach) and censoring as described in the SAP. Censored subjects were considered to be not anymore under risk for a q8 need identification at later visits. Corresponding 95% Confidence Intervals (CIs) were derived from the LOGLOG transformation. This outcome measure was pre-specified for brolucizumab 6 mg arm only. Hypothesis testing not pre-specified.
Time Frame: Weeks 16, 20, 28, 32, 40, 44, 52, 56, 64, 68, 76, 80, 88, 92, 96
Population: FAS - efficacy/safety approach
Measure: Number (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 370
proportion of subjects | 0.3856 [0.3336 to 0.4372]

6. Secondary Outcome: Proportion of Subjects With Positive q12 Treatment Status at Week 96 Within the Subjects With no q8 Treatment Need During the Initial q12w Cycle (Week 16, Week 20)
Description: as for outcome 5
Time Frame: Weeks 16, 20, 28, 32, 40, 44, 52, 56, 64, 68, 76, 80, 88, 92, 96
Population: FAS - efficacy/safety approach
Measure: Number (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 221
proportion of subjects | 0.6170 [0.5465 to 0.6799]

7. Secondary Outcome: Change From Baseline in BCVA (Letters Read) at Each Post-baseline Visit - Study Eye
Description: BCVA (with spectacles or other visual corrective devices) was assessed using ETDRS testing at 4 meters and reported in letters read correctly. Baseline was defined as the last measurement prior to first treatment. An increase (gain) in letters read from the baseline assessment indicates improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
letters
  Change from baseline at Week 4 | 3.7 (7.03) | 4.7 (7.62)
  Change from baseline at Week 8 | 5.0 (8.16) | 6.0 (9.32)
  Change from baseline at Week 12 | 5.4 (9.35) | 6.4 (10.14)
  Change from baseline at Week 16 | 5.4 (9.65) | 6.3 (10.46)
  Change from baseline at Week 20 | 5.4 (10.42) | 6.9 (10.66)
  Change from baseline at Week 24 | 5.8 (10.76) | 6.7 (11.17)
  Change from baseline at Week 28 | 6.3 (10.97) | 7.4 (11.86)
  Change from baseline at Week 32 | 6.5 (10.92) | 7.3 (11.44)
  Change from baseline at Week 36 | 6.4 (11.32) | 7.6 (11.99)
  Change from baseline at Week 40 | 6.4 (11.66) | 7.6 (11.85)
  Change from baseline at Week 44 | 6.5 (11.51) | 8.0 (12.28)
  Change from baseline at Week 48 | 6.9 (11.47) | 7.6 (12.47)
  Change from baseline at Week 52 | 6.8 (12.03) | 7.4 (12.91)
  Change from baseline at Week 56 | 6.6 (12.43) | 7.2 (13.04)
  Change from baseline at Week 60 | 6.5 (12.23) | 7.4 (13.49)
  Change from baseline at Week 64 | 6.5 (12.51) | 7.2 (13.79)
  Change from baseline at Week 68 | 6.5 (12.22) | 7.1 (14.29)
  Change from baseline at Week 72 | 6.1 (13.32) | 6.9 (13.74)
  Change from baseline at Week 76 | 6.3 (13.44) | 6.8 (13.80)
  Change from baseline at Week 80 | 6.4 (13.43) | 6.6 (13.97)
  Change from baseline at Week 84 | 5.8 (13.76) | 6.7 (14.04)
  Change from baseline at Week 88 | 6.3 (13.40) | 6.9 (14.02)
  Change from baseline at Week 92 | 6.1 (13.85) | 6.5 (14.29)
  Change from baseline at Week 96 | 6.1 (14.06) | 6.6 (14.55)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.0 to 0.0], Standard Error of Mean 0.52 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.2 to 0.2], Standard Error of Mean 0.63 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.4 to 0.4], Standard Error of Mean 0.71 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-2.3 to 0.6], Standard Error of Mean 0.73 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -1.5, 95% CI 2-sided [-3.0 to 0.0], Standard Error of Mean 0.76 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-2.5 to 0.6], Standard Error of Mean 0.79 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -1.1, 95% CI 2-sided [-2.7 to 0.5], Standard Error of Mean 0.82 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-2.5 to 0.7], Standard Error of Mean 0.81 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -1.2, 95% CI 2-sided [-2.9 to 0.4], Standard Error of Mean 0.84 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -1.2, 95% CI 2-sided [-2.9 to 0.5], Standard Error of Mean 0.85 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -1.6, 95% CI 2-sided [-3.2 to 0.1], Standard Error of Mean 0.86 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-2.4 to 1.0], Standard Error of Mean 0.86 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-2.5 to 1.1], Standard Error of Mean 0.90 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-2.5 to 1.1], Standard Error of Mean 0.92 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-2.7 to 1.0], Standard Error of Mean 0.93 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-2.5 to 1.2], Standard Error of Mean 0.95 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-2.5 to 1.2], Standard Error of Mean 0.96 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-2.8 to 1.1], Standard Error of Mean 0.98 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-2.5 to 1.4], Standard Error of Mean 0.98 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-2.1 to 1.8], Standard Error of Mean 0.99 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-2.9 to 1.1], Standard Error of Mean 1.00 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-2.6 to 1.3], Standard Error of Mean 0.99 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-2.4 to 1.6], Standard Error of Mean 1.02 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-2.5 to 1.6], Standard Error of Mean 1.04 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

8. Secondary Outcome: Average Change From Baseline in BCVA (Letters Read) Over the Period Week 4 to Week 48/96 - Study Eye
Description: as for outcome 7
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
letters
  Change from baseline over the period Week 4 to 48 | 5.8 (9.11) | 6.9 (10.11)
  Change from baseline over the period Week 4 to 96 | 6.1 (10.42) | 6.9 (11.41)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4 to Week 48; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -1.1, 95% CI 2-sided [-2.4 to 0.3], Standard Error of Mean 0.69 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4 to Week 96; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-2.4 to 0.7], Standard Error of Mean 0.78 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

9. Secondary Outcome: Average Change From Baseline in BCVA (Letters Read) Over the Period Week 12 to Week 48/96 - Study Eye
Description: as for outcome 7
Time Frame: Baseline, Weeks 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
letters
  Change from baseline over the period Week 12 to 48 | 6.1 (9.91) | 7.2 (10.77)
  Change from baseline over the period Week 12 to 96 | 6.2 (10.97) | 7.0 (11.88)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12 to Week 48; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -1.1, 95% CI 2-sided [-2.5 to 0.4], Standard Error of Mean 0.74 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12 to Week 96; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-2.4 to 0.8], Standard Error of Mean 0.82; Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

10. Secondary Outcome: Average Change From Baseline in BCVA (Letters Read) Over the Period Week 84 to Week 96 - Study Eye
Description: as for outcome 7
Time Frame: Baseline, Weeks 84, 88, 92, 96
Population: FAS - LOCF
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
letters | 6.1 (13.51) | 6.7 (13.96)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline BCVA categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-2.5 to 1.4], Standard Error of Mean 0.99 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

11. Secondary Outcome: Percentage of Subjects With >=15 Letter Gain From Baseline in BCVA (Letters Read) at Each Post-baseline Visit - Study Eye
Description: BCVA (with spectacles or other visual corrective devices) was assessed using ETDRS testing at 4 meters and reported in letters read correctly. Baseline was defined as the last measurement prior to first treatment. An increase (gain) in letters read from the baseline assessment indicates improvement. 95% confidence interval (CI) for binomial proportions was based on Clopper-Pearson exact method. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Change from baseline at Week 4 | 7.6 [5.1 to 10.8] | 8.9 [6.2 to 12.3]
  Change from baseline at Week 8 | 13.8 [10.4 to 17.7] | 18.2 [14.4 to 22.5]
  Change from baseline at Week 12 | 16.5 [12.9 to 20.7] | 21.4 [17.3 to 26.0]
  Change from baseline at Week 16 | 20.0 [16.0 to 24.4] | 22.2 [18.1 to 26.8]
  Change from baseline at Week 20 | 20.5 [16.5 to 25.0] | 23.6 [19.3 to 28.2]
  Change from baseline at Week 24 | 23.8 [19.5 to 28.5] | 22.8 [18.6 to 27.4]
  Change from baseline at Week 28 | 23.8 [19.5 to 28.5] | 27.4 [22.9 to 32.2]
  Change from baseline at Week 32 | 25.4 [21.0 to 30.2] | 28.7 [24.2 to 33.6]
  Change from baseline at Week 36 | 26.2 [21.8 to 31.0] | 30.9 [26.2 to 35.9]
  Change from baseline at Week 40 | 27.0 [22.6 to 31.9] | 31.4 [26.7 to 36.4]
  Change from baseline at Week 44 | 26.8 [22.3 to 31.6] | 31.2 [26.5 to 36.2]
  Change from baseline at Week 48 | 29.5 [24.9 to 34.4] | 29.8 [25.2 to 34.8]
  Change from baseline at Week 52 | 30.3 [25.6 to 35.2] | 30.6 [26.0 to 35.6]
  Change from baseline at Week 56 | 29.7 [25.1 to 34.7] | 30.6 [26.0 to 35.6]
  Change from baseline at Week 60 | 28.6 [24.1 to 33.5] | 30.6 [26.0 to 35.6]
  Change from baseline at Week 64 | 29.7 [25.1 to 34.7] | 30.9 [26.2 to 35.9]
  Change from baseline at Week 68 | 28.9 [24.3 to 33.8] | 32.2 [27.5 to 37.3]
  Change from baseline at Week 72 | 27.6 [23.1 to 32.4] | 31.4 [26.7 to 36.4]
  Change from baseline at Week 76 | 28.4 [23.8 to 33.3] | 30.6 [26.0 to 35.6]
  Change from baseline at Week 80 | 28.1 [23.6 to 33.0] | 30.4 [25.7 to 35.3]
  Change from baseline at Week 84 | 27.6 [23.1 to 32.4] | 31.2 [26.5 to 36.2]
  Change from baseline at Week 88 | 27.6 [23.1 to 32.4] | 33.1 [28.3 to 38.1]
  Change from baseline at Week 92 | 29.5 [24.9 to 34.4] | 30.9 [26.2 to 35.9]
  Change from baseline at Week 96 | 29.2 [24.6 to 34.1] | 31.4 [26.7 to 36.4]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.3, 95% CI 2-sided [-5.1 to 2.9] — Statistical model used logistic regression adjusting for BCVA categories, age categories, and treatment as fixed effect factors. 95% CI for difference in proportions (Brolucizumab 6mg - Aflibercept 2mg) was estimated using a bootstrap method
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -4.3, 95% CI 2-sided [-9.5 to 1.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.0, 95% CI 2-sided [-10.5 to 0.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.3, 95% CI 2-sided [-8.4 to 3.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.1, 95% CI 2-sided [-8.8 to 2.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.9, 95% CI 2-sided [-5.2 to 6.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.7, 95% CI 2-sided [-9.9 to 2.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.6, 95% CI 2-sided [-10.5 to 2.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -4.9, 95% CI 2-sided [-11.6 to 1.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -4.7, 95% CI 2-sided [-11.5 to 1.9] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -4.6, 95% CI 2-sided [-11.3 to 1.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.6, 95% CI 2-sided [-7.1 to 5.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.6, 95% CI 2-sided [-7.0 to 5.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.1, 95% CI 2-sided [-7.7 to 5.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.2, 95% CI 2-sided [-8.3 to 4.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.4, 95% CI 2-sided [-7.9 to 5.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.5, 95% CI 2-sided [-9.9 to 3.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -4.1, 95% CI 2-sided [-10.2 to 2.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.4, 95% CI 2-sided [-8.8 to 4.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.6, 95% CI 2-sided [-9.0 to 3.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.8, 95% CI 2-sided [-9.9 to 2.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.8, 95% CI 2-sided [-11.8 to 0.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.7, 95% CI 2-sided [-7.9 to 4.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.4, 95% CI 2-sided [-8.8 to 4.1] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Percentage of Subjects With >=10 Letter Gain From Baseline in BCVA (Letters Read) at Each Post-baseline Visit - Study Eye
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Change from baseline at Week 4 | 20.0 [16.0 to 24.4] | 22.2 [18.1 to 26.8]
  Change from baseline at Week 8 | 26.8 [22.3 to 31.6] | 32.8 [28.0 to 37.8]
  Change from baseline at Week 12 | 32.4 [27.7 to 37.5] | 36.0 [31.1 to 41.2]
  Change from baseline at Week 16 | 36.5 [31.6 to 41.6] | 36.9 [31.9 to 42.0]
  Change from baseline at Week 20 | 33.8 [29.0 to 38.9] | 38.2 [33.2 to 43.4]
  Change from baseline at Week 24 | 35.7 [30.8 to 40.8] | 39.3 [34.3 to 44.5]
  Change from baseline at Week 28 | 40.3 [35.2 to 45.5] | 42.5 [37.4 to 47.8]
  Change from baseline at Week 32 | 41.1 [36.0 to 46.3] | 43.4 [38.2 to 48.6]
  Change from baseline at Week 36 | 40.3 [35.2 to 45.5] | 45.5 [40.4 to 50.8]
  Change from baseline at Week 40 | 43.5 [38.4 to 48.7] | 46.3 [41.2 to 51.6]
  Change from baseline at Week 44 | 42.4 [37.3 to 47.6] | 45.3 [40.1 to 50.5]
  Change from baseline at Week 48 | 44.1 [38.9 to 49.3] | 45.8 [40.6 to 51.0]
  Change from baseline at Week 52 | 44.9 [39.7 to 50.1] | 45.8 [40.6 to 51.0]
  Change from baseline at Week 56 | 43.0 [37.9 to 48.2] | 45.5 [40.4 to 50.8]
  Change from baseline at Week 60 | 42.2 [37.1 to 47.4] | 44.7 [39.6 to 49.9]
  Change from baseline at Week 64 | 44.3 [39.2 to 49.5] | 45.8 [40.6 to 51.0]
  Change from baseline at Week 68 | 43.5 [38.4 to 48.7] | 45.0 [39.8 to 50.2]
  Change from baseline at Week 72 | 41.1 [36.0 to 46.3] | 44.4 [39.3 to 49.7]
  Change from baseline at Week 76 | 45.4 [40.3 to 50.6] | 44.7 [39.6 to 49.9]
  Change from baseline at Week 80 | 43.8 [38.7 to 49.0] | 44.2 [39.0 to 49.4]
  Change from baseline at Week 84 | 40.8 [35.8 to 46.0] | 44.2 [39.0 to 49.4]
  Change from baseline at Week 88 | 43.2 [38.1 to 48.5] | 45.5 [40.4 to 50.8]
  Change from baseline at Week 92 | 45.4 [40.3 to 50.6] | 43.4 [38.2 to 48.6]
  Change from baseline at Week 96 | 45.1 [40.0 to 50.4] | 45.0 [39.8 to 50.2]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.1, 95% CI 2-sided [-7.6 to 3.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -6.0, 95% CI 2-sided [-13.0 to 0.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.8, 95% CI 2-sided [-10.1 to 2.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.5, 95% CI 2-sided [-7.3 to 6.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -4.6, 95% CI 2-sided [-11.2 to 2.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.7, 95% CI 2-sided [-10.7 to 3.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.4, 95% CI 2-sided [-9.6 to 4.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.6, 95% CI 2-sided [-9.4 to 4.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.4, 95% CI 2-sided [-12.1 to 1.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.1, 95% CI 2-sided [-9.9 to 3.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.0, 95% CI 2-sided [-10.3 to 4.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.9, 95% CI 2-sided [-8.7 to 4.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.3, 95% CI 2-sided [-8.0 to 5.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.8, 95% CI 2-sided [-9.8 to 4.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other — Hypothesis testing not pre-specified; Regression, Logistic; Difference in proportions = -2.8, 95% CI 2-sided [-9.6 to 4.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.7, 95% CI 2-sided [-8.8 to 5.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.7, 95% CI 2-sided [-8.4 to 5.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.6, 95% CI 2-sided [-10.4 to 2.9] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.5, 95% CI 2-sided [-6.5 to 7.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.7, 95% CI 2-sided [-7.5 to 6.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.5, 95% CI 2-sided [-10.4 to 3.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.5, 95% CI 2-sided [-9.6 to 3.9] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.9, 95% CI 2-sided [-5.0 to 8.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.1, 95% CI 2-sided [-7.0 to 6.8] — [estimate comment as in outcome 11, analysis 1]

13. Secondary Outcome: Percentage of Subjects With >=5 Letter Gain From Baseline in BCVA (Letters Read) at Each Post-baseline Visit - Study Eye
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Change from baseline at Week 4 | 41.6 [36.5 to 46.8] | 45.3 [40.1 to 50.5]
  Change from baseline at Week 8 | 50.0 [44.8 to 55.2] | 53.1 [47.9 to 58.3]
  Change from baseline at Week 12 | 55.1 [49.9 to 60.3] | 58.5 [53.3 to 63.6]
  Change from baseline at Week 16 | 55.4 [50.2 to 60.5] | 56.6 [51.4 to 61.8]
  Change from baseline at Week 20 | 55.9 [50.7 to 61.1] | 61.0 [55.8 to 66.0]
  Change from baseline at Week 24 | 58.1 [52.9 to 63.2] | 61.0 [55.8 to 66.0]
  Change from baseline at Week 28 | 60.0 [54.8 to 65.0] | 65.6 [60.5 to 70.4]
  Change from baseline at Week 32 | 64.1 [58.9 to 68.9] | 65.6 [60.5 to 70.4]
  Change from baseline at Week 36 | 63.2 [58.1 to 68.2] | 65.3 [60.2 to 70.2]
  Change from baseline at Week 40 | 63.0 [57.8 to 67.9] | 64.0 [58.8 to 68.9]
  Change from baseline at Week 44 | 64.6 [59.5 to 69.5] | 65.9 [60.8 to 70.7]
  Change from baseline at Week 48 | 64.6 [59.5 to 69.5] | 64.5 [59.4 to 69.4]
  Change from baseline at Week 52 | 63.0 [57.8 to 67.9] | 65.3 [60.2 to 70.2]
  Change from baseline at Week 56 | 62.7 [57.6 to 67.6] | 64.2 [59.1 to 69.1]
  Change from baseline at Week 60 | 62.2 [57.0 to 67.1] | 62.6 [57.4 to 67.6]
  Change from baseline at Week 64 | 65.7 [60.6 to 70.5] | 63.1 [58.0 to 68.1]
  Change from baseline at Week 68 | 62.2 [57.0 to 67.1] | 63.4 [58.3 to 68.3]
  Change from baseline at Week 72 | 63.0 [57.8 to 67.9] | 61.5 [56.3 to 66.5]
  Change from baseline at Week 76 | 63.8 [58.7 to 68.7] | 61.5 [56.3 to 66.5]
  Change from baseline at Week 80 | 65.1 [60.0 to 70.0] | 60.7 [55.5 to 65.7]
  Change from baseline at Week 84 | 61.9 [56.7 to 66.9] | 64.2 [59.1 to 69.1]
  Change from baseline at Week 88 | 63.2 [58.1 to 68.2] | 62.1 [56.9 to 67.0]
  Change from baseline at Week 92 | 64.6 [59.5 to 69.5] | 60.7 [55.5 to 65.7]
  Change from baseline at Week 96 | 64.1 [58.9 to 68.9] | 60.7 [55.5 to 65.7]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.5, 95% CI 2-sided [-10.4 to 3.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.2, 95% CI 2-sided [-10.2 to 3.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.7, 95% CI 2-sided [-10.7 to 3.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.4, 95% CI 2-sided [-8.4 to 5.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.3, 95% CI 2-sided [-12.3 to 1.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.2, 95% CI 2-sided [-9.9 to 3.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.9, 95% CI 2-sided [-12.8 to 0.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.9, 95% CI 2-sided [-8.2 to 4.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.3, 95% CI 2-sided [-9.2 to 4.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.3, 95% CI 2-sided [-8.2 to 5.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.5, 95% CI 2-sided [-8.5 to 5.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.2, 95% CI 2-sided [-7.4 to 6.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.7, 95% CI 2-sided [-9.8 to 4.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.7, 95% CI 2-sided [-8.6 to 4.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.7, 95% CI 2-sided [-7.8 to 6.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 2.3, 95% CI 2-sided [-4.5 to 9.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.5, 95% CI 2-sided [-8.6 to 4.9] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.1, 95% CI 2-sided [-5.8 to 7.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 2.0, 95% CI 2-sided [-5.1 to 8.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 4.2, 95% CI 2-sided [-2.8 to 10.9] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.7, 95% CI 2-sided [-9.3 to 4.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.9, 95% CI 2-sided [-6.1 to 7.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 3.7, 95% CI 2-sided [-3.0 to 10.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 3.1, 95% CI 2-sided [-3.9 to 10.0] — [estimate comment as in outcome 11, analysis 1]

14. Secondary Outcome: Percentage of Subjects With >=15 Letter Loss From Baseline in BCVA (Letters Read) at Each Post-baseline Visit - Study Eye
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Change from baseline at Week 4 | 1.1 [0.3 to 2.7] | 1.1 [0.3 to 2.8]
  Change from baseline at Week 8 | 1.1 [0.3 to 2.7] | 1.6 [0.6 to 3.5]
  Change from baseline at Week 12 | 1.9 [0.8 to 3.9] | 1.9 [0.8 to 3.9]
  Change from baseline at Week 16 | 2.2 [0.9 to 4.2] | 2.2 [0.9 to 4.2]
  Change from baseline at Week 20 | 3.5 [1.9 to 5.9] | 3.0 [1.5 to 5.3]
  Change from baseline at Week 24 | 2.7 [1.3 to 4.9] | 3.3 [1.7 to 5.6]
  Change from baseline at Week 28 | 3.0 [1.5 to 5.3] | 3.5 [1.9 to 5.9]
  Change from baseline at Week 32 | 3.2 [1.7 to 5.6] | 3.8 [2.1 to 6.3]
  Change from baseline at Week 36 | 3.8 [2.1 to 6.3] | 3.5 [1.9 to 5.9]
  Change from baseline at Week 40 | 5.4 [3.3 to 8.2] | 4.3 [2.5 to 6.9]
  Change from baseline at Week 44 | 4.6 [2.7 to 7.3] | 4.6 [2.7 to 7.3]
  Change from baseline at Week 48 | 3.8 [2.1 to 6.3] | 4.9 [2.9 to 7.6]
  Change from baseline at Week 52 | 4.6 [2.7 to 7.3] | 5.7 [3.6 to 8.6]
  Change from baseline at Week 56 | 5.9 [3.8 to 8.9] | 5.4 [3.3 to 8.2]
  Change from baseline at Week 60 | 6.2 [4.0 to 9.2] | 5.7 [3.6 to 8.6]
  Change from baseline at Week 64 | 6.8 [4.4 to 9.8] | 6.2 [4.0 to 9.2]
  Change from baseline at Week 68 | 5.4 [3.3 to 8.2] | 6.5 [4.2 to 9.5]
  Change from baseline at Week 72 | 7.3 [4.9 to 10.4] | 6.5 [4.2 to 9.5]
  Change from baseline at Week 76 | 6.8 [4.4 to 9.8] | 6.2 [4.0 to 9.2]
  Change from baseline at Week 80 | 7.0 [4.6 to 10.1] | 6.2 [4.0 to 9.2]
  Change from baseline at Week 84 | 7.3 [4.9 to 10.4] | 7.3 [4.9 to 10.5]
  Change from baseline at Week 88 | 6.8 [4.4 to 9.8] | 7.0 [4.7 to 10.2]
  Change from baseline at Week 92 | 7.0 [4.6 to 10.1] | 7.6 [5.1 to 10.8]
  Change from baseline at Week 96 | 7.0 [4.6 to 10.1] | 7.6 [5.1 to 10.8]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.0, 95% CI 2-sided [-1.6 to 1.4] — Statistical model used logistic regression adjusting for baseline fluid status, age categories, and treatment as fixed effect factors. 95% CI for difference in proportions (Brolucizumab 6mg - Aflibercept 2mg) was estimated using a bootstrap method
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.6, 95% CI 2-sided [-2.3 to 1.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.0, 95% CI 2-sided [-1.9 to 2.2] — Statistical model used logistic regression adjusting for BCVA categories, age categories, and treatment as fixed effect factors. 95% CI for difference in proportions (Brolucizumab 6mg - Aflibercept 2 mg) was estimated using a bootstrap method
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.0, 95% CI 2-sided [-2.1 to 2.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.6, 95% CI 2-sided [-2.0 to 3.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.5, 95% CI 2-sided [-3.0 to 2.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.5, 95% CI 2-sided [-3.0 to 2.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.5, 95% CI 2-sided [-3.2 to 2.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.4, 95% CI 2-sided [-2.3 to 3.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.2, 95% CI 2-sided [-1.7 to 4.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.1, 95% CI 2-sided [-2.7 to 3.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.0, 95% CI 2-sided [-3.9 to 2.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.0, 95% CI 2-sided [-4.3 to 2.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.6, 95% CI 2-sided [-2.8 to 3.9] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.6, 95% CI 2-sided [-2.5 to 4.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.7, 95% CI 2-sided [-2.7 to 4.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.9, 95% CI 2-sided [-4.2 to 2.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.9, 95% CI 2-sided [-2.5 to 4.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.7, 95% CI 2-sided [-2.5 to 4.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.9, 95% CI 2-sided [-2.4 to 4.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.2, 95% CI 2-sided [-3.1 to 4.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.2, 95% CI 2-sided [-3.5 to 3.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.4, 95% CI 2-sided [-3.8 to 3.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.4, 95% CI 2-sided [-3.8 to 3.3] — [estimate comment as in outcome 11, analysis 1]

15. Secondary Outcome: Percentage of Subjects With >=10 Letter Loss From Baseline in BCVA (Letters Read) at Each Post-baseline Visit - Study Eye
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Change from baseline at Week 4 | 1.9 [0.8 to 3.9] | 2.4 [1.1 to 4.6]
  Change from baseline at Week 8 | 2.2 [0.9 to 4.2] | 2.2 [0.9 to 4.2]
  Change from baseline at Week 12 | 2.7 [1.3 to 4.9] | 3.0 [1.5 to 5.3]
  Change from baseline at Week 16 | 3.8 [2.1 to 6.3] | 5.1 [3.1 to 7.9]
  Change from baseline at Week 20 | 5.9 [3.8 to 8.9] | 4.6 [2.7 to 7.3]
  Change from baseline at Week 24 | 5.1 [3.1 to 7.9] | 6.0 [3.8 to 8.9]
  Change from baseline at Week 28 | 5.9 [3.8 to 8.9] | 5.7 [3.6 to 8.6]
  Change from baseline at Week 32 | 5.9 [3.8 to 8.9] | 6.2 [4.0 to 9.2]
  Change from baseline at Week 36 | 6.5 [4.2 to 9.5] | 6.2 [4.0 to 9.2]
  Change from baseline at Week 40 | 7.0 [4.6 to 10.1] | 6.0 [3.8 to 8.9]
  Change from baseline at Week 44 | 8.6 [6.0 to 12.0] | 6.2 [4.0 to 9.2]
  Change from baseline at Week 48 | 6.8 [4.4 to 9.8] | 7.3 [4.9 to 10.5]
  Change from baseline at Week 52 | 8.1 [5.5 to 11.4] | 7.3 [4.9 to 10.5]
  Change from baseline at Week 56 | 9.2 [6.4 to 12.6] | 8.1 [5.6 to 11.4]
  Change from baseline at Week 60 | 8.1 [5.5 to 11.4] | 7.3 [4.9 to 10.5]
  Change from baseline at Week 64 | 8.4 [5.8 to 11.7] | 8.7 [6.0 to 12.0]
  Change from baseline at Week 68 | 7.6 [5.1 to 10.8] | 8.4 [5.8 to 11.7]
  Change from baseline at Week 72 | 7.8 [5.3 to 11.1] | 8.1 [5.6 to 11.4]
  Change from baseline at Week 76 | 9.5 [6.7 to 12.9] | 9.2 [6.5 to 12.6]
  Change from baseline at Week 80 | 9.2 [6.4 to 12.6] | 10.0 [7.2 to 13.6]
  Change from baseline at Week 84 | 9.5 [6.7 to 12.9] | 9.5 [6.7 to 12.9]
  Change from baseline at Week 88 | 8.9 [6.2 to 12.3] | 9.8 [6.9 to 13.3]
  Change from baseline at Week 92 | 9.2 [6.4 to 12.6] | 11.1 [8.1 to 14.8]
  Change from baseline at Week 96 | 9.2 [6.4 to 12.6] | 10.3 [7.4 to 13.9]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.5, 95% CI 2-sided [-2.6 to 1.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.0, 95% CI 2-sided [-2.2 to 2.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.3, 95% CI 2-sided [-2.8 to 2.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.4, 95% CI 2-sided [-4.4 to 1.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.4, 95% CI 2-sided [-1.7 to 4.9] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.7, 95% CI 2-sided [-3.9 to 2.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.3, 95% CI 2-sided [-3.2 to 3.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.1, 95% CI 2-sided [-3.8 to 3.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.3, 95% CI 2-sided [-3.0 to 4.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.2, 95% CI 2-sided [-2.4 to 5.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 2.5, 95% CI 2-sided [-1.1 to 6.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.4, 95% CI 2-sided [-4.0 to 3.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.9, 95% CI 2-sided [-2.8 to 4.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.2, 95% CI 2-sided [-2.8 to 5.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference of proportions = 1.0, 95% CI 2-sided [-2.6 to 4.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.1, 95% CI 2-sided [-4.0 to 4.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.6, 95% CI 2-sided [-4.2 to 3.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.1, 95% CI 2-sided [-4.0 to 3.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.4, 95% CI 2-sided [-3.5 to 4.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.7, 95% CI 2-sided [-4.5 to 3.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.2, 95% CI 2-sided [-3.6 to 4.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.7, 95% CI 2-sided [-4.5 to 3.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.8, 95% CI 2-sided [-5.7 to 2.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.0, 95% CI 2-sided [-4.9 to 3.2] — [estimate comment as in outcome 11, analysis 1]

16. Secondary Outcome: Percentage of Subjects With >=5 Letter Loss From Baseline in BCVA (Letters Read) at Each Post-baseline Visit - Study Eye
Description: as for outcome 11
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Change from baseline at Week 4 | 6.2 [4.0 to 9.2] | 6.5 [4.2 to 9.5]
  Change from baseline at Week 8 | 7.8 [5.3 to 11.1] | 8.4 [5.8 to 11.7]
  Change from baseline at Week 12 | 8.4 [5.8 to 11.7] | 9.5 [6.7 to 12.9]
  Change from baseline at Week 16 | 10.8 [7.8 to 14.4] | 8.9 [6.2 to 12.3]
  Change from baseline at Week 20 | 11.6 [8.5 to 15.3] | 8.1 [5.6 to 11.4]
  Change from baseline at Week 24 | 13.0 [9.7 to 16.8] | 10.0 [7.2 to 13.6]
  Change from baseline at Week 28 | 11.4 [8.3 to 15.0] | 8.9 [6.2 to 12.3]
  Change from baseline at Week 32 | 12.2 [9.0 to 15.9] | 11.1 [8.1 to 14.8]
  Change from baseline at Week 36 | 12.7 [9.5 to 16.5] | 9.5 [6.7 to 12.9]
  Change from baseline at Week 40 | 11.9 [8.8 to 15.6] | 11.1 [8.1 to 14.8]
  Change from baseline at Week 44 | 11.9 [8.8 to 15.6] | 9.2 [6.5 to 12.6]
  Change from baseline at Week 48 | 11.1 [8.1 to 14.7] | 11.9 [8.8 to 15.7]
  Change from baseline at Week 52 | 13.2 [10.0 to 17.1] | 11.4 [8.3 to 15.1]
  Change from baseline at Week 56 | 13.2 [10.0 to 17.1] | 11.7 [8.6 to 15.4]
  Change from baseline at Week 60 | 12.7 [9.5 to 16.5] | 11.7 [8.6 to 15.4]
  Change from baseline at Week 64 | 12.7 [9.5 to 16.5] | 12.5 [9.3 to 16.3]
  Change from baseline at Week 68 | 13.8 [10.4 to 17.7] | 12.2 [9.0 to 16.0]
  Change from baseline at Week 72 | 14.1 [10.7 to 18.0] | 13.6 [10.2 to 17.5]
  Change from baseline at Week 76 | 14.1 [10.7 to 18.0] | 13.6 [10.2 to 17.5]
  Change from baseline at Week 80 | 13.8 [10.4 to 17.7] | 15.2 [11.7 to 19.3]
  Change from baseline at Week 84 | 14.1 [10.7 to 18.0] | 14.6 [11.2 to 18.7]
  Change from baseline at Week 88 | 13.0 [9.7 to 16.8] | 14.4 [10.9 to 18.4]
  Change from baseline at Week 92 | 14.3 [10.9 to 18.3] | 16.0 [12.4 to 20.1]
  Change from baseline at Week 96 | 14.3 [10.9 to 18.3] | 14.6 [11.2 to 18.7]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.2, 95% CI 2-sided [-3.5 to 3.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.5, 95% CI 2-sided [-4.4 to 3.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.0, 95% CI 2-sided [-5.0 to 3.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.9, 95% CI 2-sided [-1.9 to 6.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 3.7, 95% CI 2-sided [-0.4 to 7.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Number of subjects with >=5 letter loss from baseline in BCVA (letters read) at each post-baseline visit - Week 24; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 3.1, 95% CI 2-sided [-1.3 to 7.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 2.6, 95% CI 2-sided [-1.7 to 7.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.2, 95% CI 2-sided [-3.2 to 5.9] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 3.4, 95% CI 2-sided [-0.7 to 8.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.0, 95% CI 2-sided [-3.8 to 5.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 2.9, 95% CI 2-sided [-1.4 to 7.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.7, 95% CI 2-sided [-5.1 to 3.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 2.1, 95% CI 2-sided [-2.5 to 6.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.8, 95% CI 2-sided [-2.8 to 6.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.2, 95% CI 2-sided [-3.6 to 5.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.5, 95% CI 2-sided [-4.0 to 5.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.8, 95% CI 2-sided [-2.8 to 6.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.7, 95% CI 2-sided [-4.3 to 5.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.7, 95% CI 2-sided [-4.4 to 5.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.2, 95% CI 2-sided [-6.0 to 3.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.4, 95% CI 2-sided [-5.2 to 4.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.2, 95% CI 2-sided [-5.7 to 3.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.5, 95% CI 2-sided [-6.5 to 3.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.1, 95% CI 2-sided [-5.1 to 4.8] — [estimate comment as in outcome 11, analysis 1]

17. Secondary Outcome: Percentage of Subjects With BCVA of 73 Letters Read or More at Each Visit - Study Eye
Description: BCVA (with spectacles or other visual corrective devices) was assessed using ETDRS testing at 4 meters and reported in letters read correctly (0-100 letters). A score of 65 to 70 letters represents a low to moderate visual acuity. Baseline was defined as the last measurement prior to first treatment. 95% confidence interval (CI) for binomial proportions was based on Clopper-Pearson exact method. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Baseline | 21.4 [17.3 to 25.9] | 17.9 [14.1 to 22.2]
  Week 4 | 31.9 [27.2 to 36.9] | 34.7 [29.8 to 39.8]
  Week 8 | 40.3 [35.2 to 45.5] | 41.2 [36.1 to 46.4]
  Week 12 | 43.5 [38.4 to 48.7] | 44.7 [39.6 to 49.9]
  Week 16 | 44.1 [38.9 to 49.3] | 42.5 [37.4 to 47.8]
  Week 20 | 44.1 [38.9 to 49.3] | 45.0 [39.8 to 50.2]
  Week 24 | 45.4 [40.3 to 50.6] | 47.4 [42.2 to 52.7]
  Week 28 | 48.6 [43.4 to 53.9] | 50.4 [45.2 to 55.6]
  Week 32 | 47.8 [42.6 to 53.1] | 49.6 [44.4 to 54.8]
  Week 36 | 47.6 [42.4 to 52.8] | 49.9 [44.6 to 55.1]
  Week 40 | 48.9 [43.7 to 54.1] | 49.3 [44.1 to 54.5]
  Week 44 | 50.3 [45.1 to 55.5] | 50.4 [45.2 to 55.6]
  Week 48 | 51.4 [46.1 to 56.6] | 49.6 [44.4 to 54.8]
  Week 52 | 49.7 [44.5 to 54.9] | 50.1 [44.9 to 55.4]
  Week 56 | 50.5 [45.3 to 55.7] | 50.9 [45.7 to 56.2]
  Week 60 | 48.9 [43.7 to 54.1] | 52.3 [47.1 to 57.5]
  Week 64 | 49.2 [44.0 to 54.4] | 50.7 [45.5 to 55.9]
  Week 68 | 48.9 [43.7 to 54.1] | 50.7 [45.5 to 55.9]
  Week 72 | 48.9 [43.7 to 54.1] | 49.3 [44.1 to 54.5]
  Week 76 | 48.9 [43.7 to 54.1] | 49.9 [44.6 to 55.1]
  Week 80 | 51.9 [46.7 to 57.1] | 50.1 [44.9 to 55.4]
  Week 84 | 48.4 [43.2 to 53.6] | 49.6 [44.4 to 54.8]
  Week 88 | 50.5 [45.3 to 55.7] | 50.7 [45.5 to 55.9]
  Week 92 | 50.5 [45.3 to 55.7] | 49.9 [44.6 to 55.1]
  Week 96 | 48.1 [42.9 to 53.3] | 49.1 [43.8 to 54.3]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -4.0, 95% CI 2-sided [-9.2 to 1.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.1, 95% CI 2-sided [-8.1 to 3.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.5, 95% CI 2-sided [-8.4 to 3.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.3, 95% CI 2-sided [-5.4 to 6.7] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.2, 95% CI 2-sided [-8.2 to 4.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.1, 95% CI 2-sided [-9.0 to 3.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.2, 95% CI 2-sided [-9.3 to 2.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.1, 95% CI 2-sided [-9.6 to 2.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.7, 95% CI 2-sided [-9.6 to 2.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.7, 95% CI 2-sided [-7.6 to 4.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.4, 95% CI 2-sided [-7.5 to 5.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.4, 95% CI 2-sided [-5.4 to 6.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.8, 95% CI 2-sided [-7.7 to 4.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.9, 95% CI 2-sided [-7.7 to 4.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -4.7, 95% CI 2-sided [-10.8 to 1.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.8, 95% CI 2-sided [-8.9 to 3.2] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.1, 95% CI 2-sided [-9.5 to 2.9] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.6, 95% CI 2-sided [-7.9 to 4.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.0, 95% CI 2-sided [-8.1 to 4.1] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.5, 95% CI 2-sided [-5.6 to 6.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.4, 95% CI 2-sided [-8.3 to 3.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.3, 95% CI 2-sided [-7.4 to 4.5] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.5, 95% CI 2-sided [-6.5 to 5.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.0, 95% CI 2-sided [-8.1 to 4.1] — [estimate comment as in outcome 11, analysis 1]

18. Secondary Outcome: Change From Baseline in Central Subfield Thickness (CSFT) at Each Post-baseline Visit - Study Eye
Description: CSFT (the average retinal thickness of the circular area within 1 millimeter diameter around the foveal center) was assessed using Spectral-Domain Optical Coherence Tomography (SD-OCT), a non-invasive measurement which produces cross-sectional and 3-dimensional images of the eye. A negative change value indicates an improvement, while a positive change value indicates a worsening. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
micrometers
  Change from baseline at Week 4 | -160.7 (126.55) | -149.2 (111.60)
  Change from baseline at Week 8 | -181.8 (142.11) | -159.6 (120.93)
  Change from baseline at Week 12 | -190.5 (148.05) | -167.6 (123.66)
  Change from baseline at Week 16 | -170.9 (152.48) | -137.7 (136.76)
  Change from baseline at Week 20 | -161.0 (151.81) | -165.3 (132.70)
  Change from baseline at Week 24 | -177.8 (150.62) | -137.3 (139.32)
  Change from baseline at Week 28 | -182.7 (156.04) | -166.6 (138.22)
  Change from baseline at Week 32 | -168.9 (157.61) | -142.6 (135.87)
  Change from baseline at Week 36 | -192.6 (156.51) | -170.2 (131.42)
  Change from baseline at Week 40 | -183.4 (156.83) | -146.5 (142.69)
  Change from baseline at Week 44 | -183.8 (161.42) | -172.7 (135.06)
  Change from baseline at Week 48 | -189.8 (158.35) | -147.8 (144.97)
  Change from baseline at Week 52 | -193.8 (157.22) | -173.9 (134.84)
  Change from baseline at Week 56 | -184.9 (162.66) | -149.9 (145.37)
  Change from baseline at Week 60 | -195.4 (161.34) | -172.2 (136.58)
  Change from baseline at Week 64 | -190.9 (160.06) | -153.1 (144.45)
  Change from baseline at Week 68 | -188.4 (161.63) | -172.9 (136.76)
  Change from baseline at Week 72 | -192.3 (160.70) | -153.1 (145.02)
  Change from baseline at Week 76 | -193.1 (162.00) | -173.1 (138.96)
  Change from baseline at Week 80 | -188.2 (165.90) | -155.6 (147.09)
  Change from baseline at Week 84 | -196.2 (161.97) | -173.4 (142.11)
  Change from baseline at Week 88 | -192.7 (162.46) | -158.3 (147.24)
  Change from baseline at Week 92 | -194.9 (162.35) | -173.9 (142.30)
  Change from baseline at Week 96 | -193.6 (163.97) | -159.3 (146.26)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -17.7, 95% CI 2-sided [-32.6 to -2.9], Standard Error of Mean 7.57 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -29.5, 95% CI 2-sided [-45.6 to -13.4], Standard Error of Mean 8.18 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -30.3, 95% CI 2-sided [-46.9 to -13.7], Standard Error of Mean 8.45 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -40.2, 95% CI 2-sided [-58.9 to -21.6], Standard Error of Mean 9.51 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -2.9, 95% CI 2-sided [-20.9 to 15.0], Standard Error of Mean 9.12 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -47.8, 95% CI 2-sided [-66.3 to -29.3], Standard Error of Mean 9.42 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -23.7, 95% CI 2-sided [-42.0 to -5.4], Standard Error of Mean 9.34 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -33.7, 95% CI 2-sided [-52.4 to -15.0], Standard Error of Mean 9.54 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -30.4, 95% CI 2-sided [-48.0 to -12.9], Standard Error of Mean 8.94 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -44.7, 95% CI 2-sided [-63.5 to -25.9], Standard Error of Mean 9.57 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -19.2, 95% CI 2-sided [-37.3 to -1.1], Standard Error of Mean 9.24 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -49.9, 95% CI 2-sided [-68.9 to -30.9], Standard Error of Mean 9.68 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -28.1, 95% CI 2-sided [-45.8 to -10.4], Standard Error of Mean 9.01 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -43.1, 95% CI 2-sided [-62.4 to -23.7], Standard Error of Mean 9.86 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -31.1, 95% CI 2-sided [-49.5 to -12.8], Standard Error of Mean 9.34 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -45.8, 95% CI 2-sided [-64.9 to -26.8], Standard Error of Mean 9.70 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -23.7, 95% CI 2-sided [-42.0 to -5.4], Standard Error of Mean 9.31 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -47.3, 95% CI 2-sided [-66.4 to -28.3], Standard Error of Mean 9.69 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -28.0, 95% CI 2-sided [-46.5 to -9.5], Standard Error of Mean 9.43 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -40.9, 95% CI 2-sided [-60.4 to -21.4], Standard Error of Mean 9.94 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -31.0, 95% CI 2-sided [-49.6 to -12.4], Standard Error of Mean 9.48 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -42.6, 95% CI 2-sided [-61.9 to -23.3], Standard Error of Mean 9.84 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -29.1, 95% CI 2-sided [-47.9 to -10.3], Standard Error of Mean 9.56 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -42.6, 95% CI 2-sided [-62.0 to -23.3], Standard Error of Mean 9.87 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

19. Secondary Outcome: Average Change From Baseline in CSFT Over the Period Week 36 Through Week 48 - Study Eye
Description: CSFT (the average retinal thickness of the circular area within 1 millimeter diameter around the foveal center) was assessed using SD-OCT, a non-invasive measurement which produces cross-sectional and 3-dimensional images of the eye. A negative change value indicates an improvement, while a positive change value indicates a worsening. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Weeks 36, 40, 44, 48
Population: FAS - LOCF
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
micrometers | -187.4 (155.58) | -159.3 (135.92)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT-total categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -36.1, 95% CI 2-sided [-54.0 to -18.1], Standard Error of Mean 9.13 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

20. Secondary Outcome: Average Change From Baseline in CSFT Over the Period Week 84 Through Week 96 - Study Eye
Description: as for outcome 19
Time Frame: Baseline, Weeks 84, 88, 92, 96
Population: FAS - LOCF
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
micrometers | -194.3 (161.24) | -166.2 (142.81)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT-total categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -36.3, 95% CI 2-sided [-55.1 to -17.6], Standard Error of Mean 9.56 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

21. Secondary Outcome: Average Change From Baseline in CSFT Over the Period Week 4 Through Week 48/96 - Study Eye
Description: as for outcome 19
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
micrometers
  Change from baseline over the period Week 4 to 48 | -178.7 (145.33) | -155.3 (126.83)
  Change from baseline over the period Week 4 to 96 | -185.4 (151.35) | -159.7 (131.74)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4 to Week 48; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT-total categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -30.8, 95% CI 2-sided [-47.6 to -14.1], Standard Error of Mean 8.53 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4 to Week 96; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT-total categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -33.5, 95% CI 2-sided [-50.8 to -16.1], Standard Error of Mean 8.84 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

22. Secondary Outcome: Change From Baseline in Choroidal Neovascularization (CNV) Lesion Size at Week 12, Week 48, and Week 96 - Study Eye
Description: CNV lesion size (the area of new blood vessels in the choroid layer of the retina) size was measured using fluorescein angiography (FA). A negative change value indicates a reduction in lesion size, whereas a positive change value indicates an increase. An increase in CNV lesion size may indicate progression of the underlying disease. Only one eye (study eye) contributed to the analysis.
Time Frame: Baseline, Weeks 12, 48, 96
Population: FAS - LOCF
Measure: Mean (Standard Deviation); unit: millimeters squared
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
millimeters squared
  Change from baseline at Week 12 | -2.2 (2.71) | -2.5 (4.02)
  Change from baseline at Week 48 | -2.3 (2.76) | -2.5 (4.04)
  Change from baseline at Week 96 | -2.5 (2.77) | -2.7 (4.03)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline lesion size categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = 0.3, 95% CI 2-sided [0.0 to 0.7], Standard Error of Mean 0.18 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline lesion size categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.6], Standard Error of Mean 0.17 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline lesion size categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = 0.3, 95% CI 2-sided [0.0 to 0.6], Standard Error of Mean 0.16 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

23. Secondary Outcome: Change From Baseline in Central Subfield Neurosensory Retinal Thickness (CSFTns) at Each Post-baseline Visit - Study Eye
Description: CSFTns was assessed using SD-OCT. A negative change value indicates an improvement, while a positive change value indicates a worsening. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
micrometers
  Change from baseline at Week 4 | -51.7 (91.79) | -44.2 (80.37)
  Change from baseline at Week 8 | -55.0 (94.92) | -45.4 (84.99)
  Change from baseline at Week 12 | -52.7 (96.89) | -42.4 (85.48)
  Change from baseline at Week 16 | -50.5 (98.30) | -41.2 (84.78)
  Change from baseline at Week 20 | -49.2 (95.87) | -48.1 (88.08)
  Change from baseline at Week 24 | -53.4 (98.35) | -41.8 (90.17)
  Change from baseline at Week 28 | -56.4 (99.86) | -47.3 (87.90)
  Change from baseline at Week 32 | -49.8 (99.41) | -42.0 (90.50)
  Change from baseline at Week 36 | -59.1 (101.18) | -47.8 (89.64)
  Change from baseline at Week 40 | -55.9 (100.01) | -43.2 (91.94)
  Change from baseline at Week 44 | -56.2 (106.65) | -47.1 (90.03)
  Change from baseline at Week 48 | -54.8 (100.28) | -41.8 (93.99)
  Change from baseline at Week 52 | -58.4 (102.35) | -49.1 (90.31)
  Change from baseline at Week 56 | -57.3 (100.85) | -45.8 (91.95)
  Change from baseline at Week 60 | -60.3 (100.56) | -49.3 (90.52)
  Change from baseline at Week 64 | -58.0 (100.89) | -47.5 (92.59)
  Change from baseline at Week 68 | -56.7 (100.16) | -49.5 (91.20)
  Change from baseline at Week 72 | -58.6 (101.34) | -47.3 (92.25)
  Change from baseline at Week 76 | -59.7 (101.61) | -50.2 (91.51)
  Change from baseline at Week 80 | -57.8 (102.92) | -47.6 (92.34)
  Change from baseline at Week 84 | -60.4 (102.80) | -50.6 (92.57)
  Change from baseline at Week 88 | -59.7 (101.97) | -49.1 (94.52)
  Change from baseline at Week 92 | -60.1 (102.00) | -51.0 (91.79)
  Change from baseline at Week 96 | -58.9 (102.48) | -49.4 (94.86)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; Analyzed using ANOVA model with baseline CSFT-neurosensory retina categories, age categories, and treatment as fixed effect factors; Least Squares Mean Difference = -2.1, 95% CI 2-sided [-11.6 to 7.3], Standard Error of Mean 4.80 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -3.8, 95% CI 2-sided [-13.6 to 6.0], Standard Error of Mean 4.98 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -4.5, 95% CI 2-sided [-14.3 to 5.3], Standard Error of Mean 4.98 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -3.7, 95% CI 2-sided [-13.7 to 6.4], Standard Error of Mean 5.12 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = 4.6, 95% CI 2-sided [-5.5 to 14.6], Standard Error of Mean 5.11 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -5.8, 95% CI 2-sided [-16.3 to 4.7], Standard Error of Mean 5.35 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -3.1, 95% CI 2-sided [-13.1 to 7.0], Standard Error of Mean 5.13 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-12.6 to 8.5], Standard Error of Mean 5.37 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-15.2 to 5.1], Standard Error of Mean 5.15 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -6.6, 95% CI 2-sided [-17.0 to 3.8], Standard Error of Mean 5.30 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -2.8, 95% CI 2-sided [-13.4 to 7.9], Standard Error of Mean 5.42 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-17.6 to 3.7], Standard Error of Mean 5.40 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -2.7, 95% CI 2-sided [-12.9 to 7.5], Standard Error of Mean 5.19 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-15.4 to 5.4], Standard Error of Mean 5.31 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -4.2, 95% CI 2-sided [-14.3 to 5.9], Standard Error of Mean 5.15 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -3.9, 95% CI 2-sided [-14.2 to 6.4], Standard Error of Mean 5.24 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-10.7 to 9.6], Standard Error of Mean 5.17 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -4.6, 95% CI 2-sided [-14.8 to 5.7], Standard Error of Mean 5.24 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -2.8, 95% CI 2-sided [-13.1 to 7.4], Standard Error of Mean 5.23 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -3.7, 95% CI 2-sided [-14.1 to 6.8], Standard Error of Mean 5.33 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -3.1, 95% CI 2-sided [-13.5 to 7.3], Standard Error of Mean 5.30 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-14.6 to 6.5], Standard Error of Mean 5.39 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other — Treatment difference; ANOVA; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -2.3, 95% CI 2-sided [-12.6 to 8.0], Standard Error of Mean 5.25 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other — Treatment difference; ANOVA — Hypothesis testing not pre-specified; [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-13.6 to 7.7], Standard Error of Mean 5.42 — Least squares mean difference (Brolucizumab 6mg - Aflibercept 2mg)

24. Secondary Outcome: Percentage of Subjects With Presence of Subretinal Fluid at Each Post-baseline Visit - Study Eye
Description: Subretinal fluid was assessed using SD-OCT and recorded as Present/Absent. The presence of subretinal fluid is an indicator of underlying disease. One eye (study eye) contributed to the analysis.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Week 4 | 29.2 [24.6 to 34.1] | 36.9 [31.9 to 42.0]
  Week 8 | 14.1 [10.7 to 18.0] | 22.8 [18.6 to 27.4]
  Week 12 | 13.5 [10.2 to 17.4] | 20.6 [16.6 to 25.1]
  Week 16 | 21.1 [17.0 to 25.6] | 35.5 [30.6 to 40.6]
  Week 20 | 25.1 [20.8 to 29.9] | 22.5 [18.3 to 27.1]
  Week 24 | 17.3 [13.6 to 21.5] | 36.9 [31.9 to 42.0]
  Week 28 | 15.9 [12.4 to 20.1] | 22.0 [17.8 to 26.5]
  Week 32 | 24.1 [19.8 to 28.7] | 34.4 [29.6 to 39.5]
  Week 36 | 13.5 [10.2 to 17.4] | 21.7 [17.6 to 26.2]
  Week 40 | 18.1 [14.3 to 22.4] | 33.9 [29.1 to 39.0]
  Week 44 | 23.8 [19.5 to 28.5] | 21.7 [17.6 to 26.2]
  Week 48 | 17.6 [13.8 to 21.8] | 33.9 [29.1 to 39.0]
  Week 52 | 19.7 [15.8 to 24.2] | 22.8 [18.6 to 27.4]
  Week 56 | 24.3 [20.0 to 29.0] | 33.6 [28.8 to 38.7]
  Week 60 | 20.0 [16.0 to 24.4] | 24.4 [20.1 to 29.1]
  Week 64 | 20.3 [16.3 to 24.7] | 35.5 [30.6 to 40.6]
  Week 68 | 23.2 [19.0 to 27.9] | 23.6 [19.3 to 28.2]
  Week 72 | 17.8 [14.1 to 22.1] | 34.7 [29.8 to 39.8]
  Week 76 | 21.6 [17.5 to 26.2] | 23.0 [18.8 to 27.7]
  Week 80 | 22.7 [18.5 to 27.3] | 33.9 [29.1 to 39.0]
  Week 84 | 18.9 [15.1 to 23.3] | 24.7 [20.3 to 29.4]
  Week 88 | 19.7 [15.8 to 24.2] | 31.7 [27.0 to 36.7]
  Week 92 | 17.3 [13.6 to 21.5] | 22.8 [18.6 to 27.4]
  Week 96 | 15.7 [12.1 to 19.8] | 30.4 [25.7 to 35.3]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -6.6, 95% CI 2-sided [-13.2 to -0.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -8.5, 95% CI 2-sided [-13.8 to -3.0] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -6.9, 95% CI 2-sided [-12.2 to -1.7] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -14.2, 95% CI 2-sided [-20.8 to -8.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 3.1, 95% CI 2-sided [-2.9 to 9.6] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -19.2, 95% CI 2-sided [-25.5 to -13.0] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.9, 95% CI 2-sided [-11.6 to -0.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -9.8, 95% CI 2-sided [-16.5 to -3.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -8.0, 95% CI 2-sided [-13.6 to -2.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -15.4, 95% CI 2-sided [-21.5 to -9.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 2.5, 95% CI 2-sided [-3.2 to 8.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -15.9, 95% CI 2-sided [-22.4 to -10.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.7, 95% CI 2-sided [-8.5 to 3.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other; Regression, Logistic; Hypothesis testing not pre-specified; Difference in proportions = -9.0, 95% CI 2-sided [-15.7 to -2.9] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.9, 95% CI 2-sided [-9.8 to 2.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -15.1, 95% CI 2-sided [-21.3 to -8.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.1, 95% CI 2-sided [-6.1 to 6.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -16.6, 95% CI 2-sided [-22.6 to -10.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.1, 95% CI 2-sided [-7.0 to 5.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -11.0, 95% CI 2-sided [-17.4 to -5.0] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.3, 95% CI 2-sided [-11.3 to 0.7] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -12.0, 95% CI 2-sided [-18.9 to -5.9] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.5, 95% CI 2-sided [-11.4 to 0.0] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -14.5, 95% CI 2-sided [-20.3 to -8.3] — [estimate comment as in outcome 14, analysis 1]

25. Secondary Outcome: Percentage of Subjects With Presence of Intraretinal Fluid at Each Post-baseline Visit - Study Eye
Description: Intraretinal fluid was assessed using SD-OCT and recorded as Present/Absent. The presence of intraretinal fluid is an indicator of underlying disease. One eye (study eye) contributed to the analysis.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Week 4 | 10.3 [7.4 to 13.8] | 8.4 [5.8 to 11.7]
  Week 8 | 7.0 [4.6 to 10.1] | 8.7 [6.0 to 12.0]
  Week 12 | 7.6 [5.1 to 10.8] | 8.7 [6.0 to 12.0]
  Week 16 | 12.7 [9.5 to 16.5] | 11.9 [8.8 to 15.7]
  Week 20 | 16.5 [12.9 to 20.7] | 7.9 [5.3 to 11.1]
  Week 24 | 10.5 [7.6 to 14.1] | 13.0 [9.7 to 16.9]
  Week 28 | 9.2 [6.4 to 12.6] | 6.0 [3.8 to 8.9]
  Week 32 | 14.3 [10.9 to 18.3] | 14.1 [10.7 to 18.1]
  Week 36 | 7.0 [4.6 to 10.1] | 8.4 [5.8 to 11.7]
  Week 40 | 13.2 [10.0 to 17.1] | 13.8 [10.5 to 17.8]
  Week 44 | 12.4 [9.2 to 16.2] | 8.1 [5.6 to 11.4]
  Week 48 | 11.1 [8.1 to 14.7] | 12.5 [9.3 to 16.3]
  Week 52 | 9.2 [6.4 to 12.6] | 7.6 [5.1 to 10.8]
  Week 56 | 13.0 [9.7 to 16.8] | 13.6 [10.2 to 17.5]
  Week 60 | 8.4 [5.8 to 11.7] | 8.4 [5.8 to 11.7]
  Week 64 | 10.3 [7.4 to 13.8] | 11.7 [8.6 to 15.4]
  Week 68 | 11.1 [8.1 to 14.7] | 8.1 [5.6 to 11.4]
  Week 72 | 11.1 [8.1 to 14.7] | 10.6 [7.6 to 14.2]
  Week 76 | 9.2 [6.4 to 12.6] | 8.4 [5.8 to 11.7]
  Week 80 | 12.4 [9.2 to 16.2] | 12.2 [9.0 to 16.0]
  Week 84 | 10.5 [7.6 to 14.1] | 9.2 [6.5 to 12.6]
  Week 88 | 10.8 [7.8 to 14.4] | 10.6 [7.6 to 14.2]
  Week 92 | 10.8 [7.8 to 14.4] | 6.8 [4.4 to 9.8]
  Week 96 | 10.8 [7.8 to 14.4] | 10.3 [7.4 to 13.9]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.5, 95% CI 2-sided [-2.5 to 5.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.1, 95% CI 2-sided [-6.1 to 1.7] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.4, 95% CI 2-sided [-5.3 to 2.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.1, 95% CI 2-sided [-4.5 to 4.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 8.2, 95% CI 2-sided [3.9 to 12.8] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.2, 95% CI 2-sided [-7.9 to 1.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 2.8, 95% CI 2-sided [-1.0 to 6.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.5, 95% CI 2-sided [-5.5 to 4.0] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.8, 95% CI 2-sided [-5.6 to 1.8] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.3, 95% CI 2-sided [-6.0 to 3.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 3.8, 95% CI 2-sided [-0.5 to 8.0] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.0, 95% CI 2-sided [-6.2 to 2.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.2, 95% CI 2-sided [-2.5 to 5.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.2, 95% CI 2-sided [-5.9 to 3.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.6, 95% CI 2-sided [-4.4 to 3.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.8, 95% CI 2-sided [-6.2 to 2.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 2.6, 95% CI 2-sided [-1.2 to 6.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.2, 95% CI 2-sided [-4.2 to 4.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.4, 95% CI 2-sided [-3.5 to 4.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.3, 95% CI 2-sided [-4.8 to 4.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.9, 95% CI 2-sided [-3.3 to 5.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.1, 95% CI 2-sided [-4.5 to 3.9] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 3.8, 95% CI 2-sided [-0.1 to 8.0] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.2, 95% CI 2-sided [-4.3 to 4.6] — [estimate comment as in outcome 14, analysis 1]

26. Secondary Outcome: Percentage of Subjects With Presence of Sub-retinal Pigment Epithelium (RPE) Fluid at Each Post-baseline Visit - Study Eye
Description: Sub-retinal pigment epithelium (RPE) fluid was assessed using SD-OCT and recorded as Present/Absent. The presence of sub-RPE fluid is an indicator of underlying disease. One eye (study eye) contributed to the analysis.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Week 4 | 18.1 [14.3 to 22.4] | 21.7 [17.6 to 26.2]
  Week 8 | 16.2 [12.6 to 20.4] | 18.7 [14.9 to 23.1]
  Week 12 | 15.9 [12.4 to 20.1] | 17.6 [13.9 to 21.9]
  Week 16 | 15.9 [12.4 to 20.1] | 23.8 [19.6 to 28.5]
  Week 20 | 17.3 [13.6 to 21.5] | 16.0 [12.4 to 20.1]
  Week 24 | 10.5 [7.6 to 14.1] | 18.4 [14.6 to 22.8]
  Week 28 | 13.8 [10.4 to 17.7] | 15.7 [12.2 to 19.8]
  Week 32 | 18.1 [14.3 to 22.4] | 23.3 [19.1 to 28.0]
  Week 36 | 13.2 [10.0 to 17.1] | 18.7 [14.9 to 23.1]
  Week 40 | 15.4 [11.9 to 19.5] | 21.4 [17.3 to 26.0]
  Week 44 | 14.9 [11.4 to 18.9] | 14.4 [10.9 to 18.4]
  Week 48 | 13.0 [9.7 to 16.8] | 22.0 [17.8 to 26.5]
  Week 52 | 17.3 [13.6 to 21.5] | 19.0 [15.1 to 23.3]
  Week 56 | 19.7 [15.8 to 24.2] | 24.9 [20.6 to 29.7]
  Week 60 | 15.9 [12.4 to 20.1] | 21.7 [17.6 to 26.2]
  Week 64 | 19.2 [15.3 to 23.6] | 24.1 [19.8 to 28.8]
  Week 68 | 18.1 [14.3 to 22.4] | 23.3 [19.1 to 28.0]
  Week 72 | 17.0 [13.3 to 21.3] | 23.8 [19.6 to 28.5]
  Week 76 | 16.5 [12.9 to 20.7] | 22.0 [17.8 to 26.5]
  Week 80 | 21.1 [17.0 to 25.6] | 27.6 [23.1 to 32.5]
  Week 84 | 23.2 [19.0 to 27.9] | 24.7 [20.3 to 29.4]
  Week 88 | 21.9 [17.8 to 26.5] | 26.8 [22.4 to 31.7]
  Week 92 | 17.3 [13.6 to 21.5] | 23.0 [18.8 to 27.7]
  Week 96 | 16.5 [12.9 to 20.7] | 22.5 [18.3 to 27.1]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.5, 95% CI 2-sided [-8.9 to 1.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.6, 95% CI 2-sided [-7.6 to 2.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.6, 95% CI 2-sided [-6.9 to 3.7] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -7.8, 95% CI 2-sided [-13.0 to -2.7] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 1.3, 95% CI 2-sided [-3.6 to 6.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -7.9, 95% CI 2-sided [-12.6 to -3.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.1, 95% CI 2-sided [-6.8 to 2.7] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.3, 95% CI 2-sided [-10.5 to -0.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.5, 95% CI 2-sided [-10.3 to -0.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -6.0, 95% CI 2-sided [-11.2 to -0.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.5, 95% CI 2-sided [-4.8 to 5.6] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -9.1, 95% CI 2-sided [-13.8 to -3.9] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.8, 95% CI 2-sided [-7.1 to 3.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.2, 95% CI 2-sided [-11.1 to 0.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.6, 95% CI 2-sided [-10.9 to -0.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.1, 95% CI 2-sided [-10.9 to 0.6] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.2, 95% CI 2-sided [-11.0 to -0.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -6.9, 95% CI 2-sided [-12.5 to -1.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.5, 95% CI 2-sided [-10.7 to -0.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -6.5, 95% CI 2-sided [-12.4 to -0.9] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -1.4, 95% CI 2-sided [-7.0 to 4.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -4.8, 95% CI 2-sided [-10.5 to 1.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.6, 95% CI 2-sided [-11.4 to 0.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.9, 95% CI 2-sided [-11.5 to -0.3] — [estimate comment as in outcome 14, analysis 1]

27. Secondary Outcome: Percentage of Subjects With Presence of Subretinal and/or Intraretinal Fluid (Central Subfield) at Each Post-baseline Visit - Study Eye
Description: Subretinal fluid and intraretinal fluid were assessed using SD-OCT and recorded as Present/Absent. The presence of subretinal and/or intraretinal fluid is an indicator of underlying disease. 95% confidence interval (CI) for binomial proportions was based on Clopper-Pearson exact method. One eye (study eye) contributed to the analysis.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96
Population: FAS - LOCF
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Week 4 | 35.9 [31.1 to 41.1] | 42.8 [37.7 to 48.0]
  Week 8 | 20.3 [16.3 to 24.7] | 29.3 [24.7 to 34.2]
  Week 12 | 19.2 [15.3 to 23.6] | 27.6 [23.1 to 32.5]
  Week 16 | 29.7 [25.1 to 34.7] | 44.7 [39.6 to 49.9]
  Week 20 | 37.8 [32.9 to 43.0] | 29.8 [25.2 to 34.8]
  Week 24 | 25.7 [21.3 to 30.4] | 45.3 [40.1 to 50.5]
  Week 28 | 23.8 [19.5 to 28.5] | 27.4 [22.9 to 32.2]
  Week 32 | 34.6 [29.8 to 39.7] | 43.9 [38.8 to 49.1]
  Week 36 | 19.5 [15.5 to 23.9] | 28.5 [23.9 to 33.4]
  Week 40 | 28.4 [23.8 to 33.3] | 44.4 [39.3 to 49.7]
  Week 44 | 33.0 [28.2 to 38.0] | 29.3 [24.7 to 34.2]
  Week 48 | 25.9 [21.6 to 30.7] | 43.6 [38.5 to 48.9]
  Week 52 | 27.0 [22.6 to 31.9] | 29.5 [24.9 to 34.5]
  Week 56 | 34.3 [29.5 to 39.4] | 43.1 [38.0 to 48.3]
  Week 60 | 26.8 [22.3 to 31.6] | 32.0 [27.2 to 37.0]
  Week 64 | 28.4 [23.8 to 33.3] | 43.4 [38.2 to 48.6]
  Week 68 | 31.9 [27.2 to 36.9] | 30.6 [26.0 to 35.6]
  Week 72 | 27.0 [22.6 to 31.9] | 41.5 [36.4 to 46.7]
  Week 76 | 29.5 [24.9 to 34.4] | 29.8 [25.2 to 34.8]
  Week 80 | 32.7 [27.9 to 37.7] | 42.5 [37.4 to 47.8]
  Week 84 | 27.3 [22.8 to 32.1] | 31.4 [26.7 to 36.4]
  Week 88 | 28.4 [23.8 to 33.3] | 38.8 [33.8 to 43.9]
  Week 92 | 25.7 [21.3 to 30.4] | 28.2 [23.6 to 33.1]
  Week 96 | 24.6 [20.3 to 29.3] | 38.2 [33.2 to 43.4]
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -6.9, 95% CI 2-sided [-14.2 to 0.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -9.2, 95% CI 2-sided [-15.5 to -2.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -8.7, 95% CI 2-sided [-15.0 to -2.6] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -15.7, 95% CI 2-sided [-22.9 to -9.0] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 7.7, 95% CI 2-sided [0.9 to 14.8] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -20.0, 95% CI 2-sided [-27.3 to -13.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.9, 95% CI 2-sided [-10.4 to 2.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -9.7, 95% CI 2-sided [-16.7 to -2.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -9.4, 95% CI 2-sided [-15.8 to -3.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -16.5, 95% CI 2-sided [-23.4 to -9.6] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 3.4, 95% CI 2-sided [-3.3 to 10.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -18.1, 95% CI 2-sided [-24.9 to -11.8] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -3.0, 95% CI 2-sided [-9.2 to 3.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 56; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -9.4, 95% CI 2-sided [-16.3 to -2.8] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 60; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -5.7, 95% CI 2-sided [-12.5 to 1.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 64; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -15.5, 95% CI 2-sided [-21.9 to -8.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 17: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 68; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = 0.9, 95% CI 2-sided [-5.9 to 7.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 72; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -14.9, 95% CI 2-sided [-21.4 to -8.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 19: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 76; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -0.8, 95% CI 2-sided [-7.5 to 5.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 80; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -10.4, 95% CI 2-sided [-17.2 to -3.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 21: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 84; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -4.5, 95% CI 2-sided [-11.4 to 2.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 88; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -11.0, 95% CI 2-sided [-18.2 to -4.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 23: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 92; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -2.9, 95% CI 2-sided [-9.4 to 3.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 96; Test type: Other; Regression, Logistic — Hypothesis testing not pre-specified; Difference in proportions = -14.1, 95% CI 2-sided [-21.3 to -7.2] — [estimate comment as in outcome 14, analysis 1]

28. Secondary Outcome: Percentage of Subjects With Disease Activity Present (q8 Treatment Need = "Yes") at Week 16 - Study Eye
Description: A disease activity assessment (DAA) was performed to identify q8 treatment need. 95% confidence interval (CI) for binomial proportions is based on Clopper-Pearson exact method. One eye (study eye) contributed to the analysis. Hypothesis testing not pre-specified.
Time Frame: Week 16
Population: FAS - 'efficacy/safety' approach. Censored data attributable to lack of efficacy and/or safety are imputed with q8w need = Yes at the next disease activity assessment visit.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects | 22.8 [18.6 to 27.5] | 32.1 [27.3 to 37.2]

29. Secondary Outcome: Change From Baseline in Visual Function Questionnaire (VFQ-25) Composite Score at Week 24, Week 48, Week 72, and Week 96
Description: The National Eye Institute Visual Function Questionnaire-25 (VFQ-25) is a validated questionnaire that collects 25 vision-targeted responses from AMD subjects. The 25 questions pertain to global vision rating (1), difficulty with near vision activities (3), difficulty with distance vision activities (3), limitations in social functioning due to vision (2), role limitations due to vision (2), dependency on others due to vision (3), mental health symptoms due to vision (4), driving difficulties (3), limitations with peripheral (1) and color vision (1), and ocular pain (2). Each response is converted to a 0 to 100 sub-scale, with the lowest and highest possible scores set at 0 and 100 points, respectively. The overall composite score (0 to 100) is obtained by averaging the 25 sub-scale scores. A high score represents better functioning.
Time Frame: Baseline, Weeks 24, 48, 72, 96
Population: FAS - Observed. Number analyzed is the number of subjects with a value for both baseline and the specific post-baseline visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
score on a scale
  Change from baseline at Week 24: number analyzed (Participants) | 354 | 355
  Change from baseline at Week 24 | 3.9 (10.09) | 3.5 (10.95)
  Change from baseline at Week 48: number analyzed (Participants) | 347 | 346
  Change from baseline at Week 48 | 4.8 (11.57) | 3.6 (11.88)
  Change from baseline at Week 72: number analyzed (Participants) | 342 | 334
  Change from baseline at Week 72 | 5.0 (13.38) | 3.2 (12.30)
  Change from baseline at Week 96: number analyzed (Participants) | 338 | 329
  Change from baseline at Week 96 | 3.8 (14.06) | 2.6 (13.11)

30. Secondary Outcome: Percentage of Subjects With Induced or Boosted Anti-drug Antibody (ADA) Status at Week 48 (Brolucizumab Only)
Description: Serum samples were collected and assessed for anti-drug antibody status. Subjects were categorized as ADA negative when one of the following was met: ADA negative at all time points (predose and postdose); ADA negative at predose and no titer values above 10 at all other time points; or ADA titer of 10 at predose but negative at all other time points. ADA induced was defined as ADA negative at predose with postdose titer value greater than or equal to a titer of 30 at any timepoint. ADA boosted was defined as ADA positive at predose with postdose titer values that increased by at least two dilutions (9-fold) from their respective predose value at any time point.
Time Frame: Week 48
Population: Safety Analysis Set - Observed
Measure: Number; unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 370
percentage of subjects | 18.8

31. Secondary Outcome: Percentage of Subjects With Intraretinal Hemorrhage (Central Subfield) Present at the Visit While Absent at Baseline at Each Treatment - Study Eye
Description: Intraretinal hemorrhage was assessed using SD-OCT and recorded as Present/Absent. The presence of intraretinal hemorrhage is an indicator of underlying disease. 95% confidence interval (CI) for binomial proportions was based on Clopper-Pearson exact method. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Weeks 12, 48, 96
Population: FAS with non-missing values. Number Analyzed represents the number of subjects with a value for both baseline and the specific post-baseline visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Week 12: number analyzed (Participants) | 260 | 290
  Week 12 | 6.9 | 6.6
  Week 48: number analyzed (Participants) | 252 | 278
  Week 48 | 4.0 | 5.0
  Week 96: number analyzed (Participants) | 242 | 260
  Week 96 | 2.1 | 2.7

32. Secondary Outcome: Percentage of Subjects With Subretinal Hemorrhage (Central Subfield) Present at the Visit While Absent at Baseline at Each Treatment - Study Eye
Description: Subretinal hemorrhage was assessed using SD-OCT and recorded as Present/Absent. The presence of subretinal hemorrhage is an indicator of underlying disease. 95% confidence interval (CI) for binomial proportions was based on Clopper-Pearson exact method. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Weeks 12, 48, 96
Population: as for outcome 31
Measure: Number; unit: percentage of subjects
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 370 | 369
percentage of subjects
  Week 12: number analyzed (Participants) | 346 | 345
  Week 12 | 0.6 | 1.2
  Week 48: number analyzed (Participants) | 333 | 329
  Week 48 | 0.6 | 0.3
  Week 96: number analyzed (Participants) | 323 | 308
  Week 96 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: First treatment through study completion, an average of 96 weeks.
Description: Adverse Events (AE) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. This analysis population includes all subjects who received at least 1 IVT injection (Safety Analysis Set).
Groups:
- Brolucizumab 6mg: All subjects exposed to brolucizumab ophthalmic solution administered as a 6 mg/50 microliter (μL) dose
- Aflibercept 2mg: All subjects exposed to aflibercept ophthalmic solution administered as a 2 mg/50 μL dose
Arm/Group | Brolucizumab 6mg | Aflibercept 2mg
All-Cause Mortality (participants affected / at risk) | 4/370 | 7/369
Serious Adverse Events (participants affected / at risk) | 79/370 | 89/369
Other Adverse Events (participants affected / at risk) | 176/370 | 194/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=370) | Aflibercept 2mg (N=369)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Parasystole (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Anterior chamber inflammation - Study eye (Eye disorders) | 1 | 0
Blindness - Study eye (Eye disorders) | 1 | 0
Dry age-related macular degeneration - Study eye (Eye disorders) | 0 | 1
Retinal artery embolism - Study eye (Eye disorders) | 1 | 0
Retinal artery occlusion - Study eye (Eye disorders) | 0 | 1
Retinal artery thrombosis - Study eye (Eye disorders) | 1 | 0
Retinal detachment - Study eye (Eye disorders) | 1 | 1
Retinal pigment epithelial tear - Study eye (Eye disorders) | 2 | 0
Retinal tear - Study eye (Eye disorders) | 2 | 1
Uveitis - Study eye (Eye disorders) | 3 | 0
Visual acuity reduced - Study eye (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lumbar hernia (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Death (General disorders) | 0 | 3
Pyrexia (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Dacryocystitis - Study eye (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endophthalmitis - Study eye (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 8
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Cataract traumatic - Study eye (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Investigation (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 4
Cerebrovascular disorder (Nervous system disorders) | 0 | 2
Ischaemic stroke (Nervous system disorders) | 2 | 1
Migraine (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Charles Bonnet syndrome (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Mental fatigue (Psychiatric disorders) | 0 | 1
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Paranoid personality disorder (Psychiatric disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Urinary bladder rupture (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hip surgery (Surgical and medical procedures) | 1 | 0
Implantable defibrillator replacement (Surgical and medical procedures) | 0 | 1
Varicose vein operation (Surgical and medical procedures) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=370) | Aflibercept 2mg (N=369)
Cataract - Fellow eye (Eye disorders) | 7 | 22
Cataract - Study eye (Eye disorders) | 11 | 43
Conjunctival haemorrhage - Study eye (Eye disorders) | 17 | 19
Eye pain - Study eye (Eye disorders) | 13 | 19
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 31 | 32
Visual acuity reduced - Study eye (Eye disorders) | 31 | 25
Bronchitis (Infections and infestations) | 22 | 20
Influenza (Infections and infestations) | 24 | 27
Nasopharyngitis (Infections and infestations) | 43 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 28
Hypertension (Vascular disorders) | 28 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT02434328/Prot_002.pdf
  • Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT02434328/SAP_001.pdf